CLINICAL TRIAL: NCT06042712
Title: Belief-updating and Speech: Potential Markers of Psychosis Relapse
Brief Title: Belief-updating, Speech and Psychosis
Acronym: BASIS
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 323994
Record Dates: First submitted 2023-09-08; First posted 2023-09-18 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Psychotic illnesses are characterised by hallucinations, delusions, and disturbed thoughts; symptoms associated with high personal and societal costs. Despite the efficacy of antipsychotic medication, approximately 84% of patients experience at least one relapse within 36 months of their first episode. Thus, identifying patients who will relapse and who will not, and then providing specific treatment to patients who are more likely to relapse is clinically meaningful. Belief-updating and speech are promising markers to predict first episode psychosis (FEP) patients future relapse outcome, as there has been evidence linking these two markers with the onset and progression of psychotic symptoms.

The present study will collect cognitive measures relating to belief-updating and speech in patients with FEP at baseline, and build models to predict relapse based on these measures. Belief updating tasks include simple video games (escaping from a planet in the Space Task and a reversal learning task). To collect speech, participants will be asked to describe ambiguous pictures. The study uses a naturalistic follow-up design; data will be collected from 140 FEP patients recruited from local clinical teams and 100 healthy controls recruited from advertisements. Cognitive tasks will be conducted via an online platform Gorilla using participants' own device (e.g. computer, laptop, smartphone and tablet). Clinical interviews can take place either online or face-to-face. Participants will attend three assessments in total, at baseline and at 6-month and 12-month follow-up. Each visit will comprise two components 1) cognitive tasks (45-60 minutes) and basic demographics, 2) clinical interviews.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria (FEP)

Participants will be recruited from two routes:

1. Participants who are part of Urban Mind study will be invited to the present study;
2. Patients who are referred to the following early psychosis teams will also be invited to the study: Lambeth Early Psychosis (LEO), Southwark Team for Early Psychosis (STEP), Lewisham Early Intervention Service (LEIS), Croydon Outreach Assessment Support Team (COAST), Central and North West London NHS Foundation Trust (NWLFT).

Participants from both routes will need to meet the following criteria:

* all participants are 18 to 40 years old
* all participants have an adequate command of the English language to complete the assessment
* all participants need access to laptop, smartphone or computer to complete the tasks
* all participants met FEP as defined by a DSM-IV diagnosis of schizophrenia, schizophreniform disorder, schizoaffective disorder, or delusional disorder based on the Structured Clinical Interview for DSM-IV (SCID-I) (First et al., 2002).

Exclusion Criteria:

Exclusion criteria (FEP)

* Experienced more than one previous episode of psychosis
* Any other neurological disorders that could potentially interfere with study process or patients' safety
* Refusing to complete the belief-updating or speech tasks
* Participants' answers are identified as fake answers or participants complete the tasks for multiple times (identified by their unique participants code).
* Participants are unable to fully comprehend the purpose of the study or make a rational decision whether or not to participate

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: People with a first episode of psychosis and matched controls
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Relapse | One year
  Change in score on the Positive and Negative Syndrome Scale